CLINICAL TRIAL: NCT01557114
Title: A Dose Escalation Phase I Study of Radiotherapy Administered in Combination With Anti-CTLA4 Monoclonal Antibody (Ipilimumab) in Patients With Unresectable Stage III or Stage IV Advanced Malignant Melanoma
Brief Title: Study of Radiotherapy Administered in Combination With Ipilimumab in Patients With Unresectable Stage III or Stage IV Advanced Malignant Melanoma
Acronym: Mel-Ipi-Rx
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: New compounds available in the indication (nivolumab/pembrolizumab), toxicity of ipilimumab
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSET 2010/1663 -Mel-Ipi-Rx; 2010-020317-93 (EudraCT Number)
Record Dates: First submitted 2011-03-16; First posted 2012-03-19 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Malignant Melanoma
Keywords: unresectable Stage III or stage IV advanced malignant melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- radiation therapy with Ipilimumab (Experimental)
  Interventions: Drug: Ipilimumab; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Ipilimumab — Induction: Treatment with ipilimumab will be administered on weeks 1, 4, 7 and 10 at 10mg/kg.
  Maintenance: Ipilimumab will be administered intravenously over 90-minutes at 10 mg/kg every 12 weeks starting at week 24, for as long as the treating physician believes that there is a clinical benefit or for as long as patient is tolerant of therapy
Radiation: Radiotherapy — Radiation therapy 9 Grays in 3 Grays fractions Radiation therapy 15 Grays in 5 Grays fractions Radiation therapy 18 Grays in 6 Grays fractions Radiation therapy 24 Grays in 8 Grays fractions

SUMMARY:
RATIONALE:Anti-melanoma activity of Ipilimumab both as a single therapy and in association with melanoma peptides has been shown as well as synergy between radiation therapy and anti-CTLA-A mAb in several tumor animal models for both local tumor control and distant effects.Radiotherapy increases tumor immunogenicity in several preclinical models by increasing MHC molecules expression and is able to induce significant tumor reduction in around 30% of cases. Thus, combining radiotherapy and administration of ipilimumab could elicit systemic antitumor response. Radiation therapy will expose tumor-associated antigens (TAA) and facilitate antigen presentation, and further blockade of CTLA-4 could amplify the immune antitumor response. In this therapeutical model, the use of the own patient tumor as a source of tumor antigens (in opposition with other vaccination protocols, where TAA are exogenic) is particularly adapted.

PURPOSE: This Phase I trial determines the side effects and best dose of radiation therapy administered in combination with ipilimumab.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary: To determine the Maximum Tolerated Dose (MTD), Dose Limiting Toxicity (DLT) and recommended Phase 2 dose of radiation therapy administered in combination with ipilimumab.

Secondary:

Adverse event profiles Preliminary anti-tumor activity following escalating doses of radiation combined to ipilimumab using the immune related response criteria irRC overall survival in patients treated with this combination systemic immunologic anti tumor response intratumoral immune response pharmacodynamic effects of ipilimumab and radiotherapy in combination on Absolute Lymphocyte Count (ALC) associations between ALC and anti-tumor activity of ipilimumab and radiotherapy in combination

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent.
* Histologic diagnosis of melanoma.
* Unresectable locally advanced or metastatic melanoma with at least one melanoma metastasis accessible to radiation therapy.
* Measurable disease according to immune related Response Criteria
* Required values for initial laboratory tests:

WBC >= 2000/uL ANC >= 1000/uL Platelets >= 75 x 103/uL Hemoglobin >= 8 g/dL Creatinine <= 2,5 x ULN AST/ALT <= 2.5 x ULN for patients without liver metastasis or <= 5 x ULN for patients with liver metastasis Total Bilirubin <= 1,5.x ULN, (except patients with Gilbert's Syndrome, who must have a total bilirubin less than 3.0 mg/dL)

* No active or chronic infection with HIV, Hepatitis B, or Hepatitis C.
* ECOG Performance status of 0 or 1.
* Men and women, >= 18 years of age.
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 8 weeks after the last dose of investigational product, in such a manner that the risk of pregnancy is minimized.

Exclusion Criteria:

* Suspected or known CNS tumors including brain metastasis.
* Any other malignancy form which the patient has been disease-free for less than 5 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix.
* Autoimmune disease: Patients with a history of inflammatory bowel disease are excluded from this study, as are patients with a history of symptomatic disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [e.g., Wegener's Granulomatosis]); motor neuropathy considered of autoimmune origin (e.g. Guillain-Barre Syndrome).
* Any underlying medical or psychiatric condition, which in the opinion of the investigator will make the administration of ipilimumab hazardous or obscure the interpretation of AEs, such as a condition associated with frequent diarrhea.
* Any non-oncology vaccine therapy used for prevention of infectious diseases (for up to 1 month before or after any dose of ipilimumab).
* A history of prior treatment with ipilimumab or prior CD137 agonist or CTLA-4 inhibitor or agonist.
* Concomitant hormonal treatment, chemotherapy or immunotherapy.
* Other investigational therapy.
* Prior radiotherapy within the same body area.
* Prior radiotherapy targeting fields containing flat bones.
* Women of childbearing potential (WOCBP), defined above
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious) illness.
* Persons of reproductive potential must agree to use an adequate method of contraception throughout treatment and for at least 8 weeks after ipilimumab is stopped.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-03; Primary Completion 2015-11 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose of radiation therapy administered in combination with ipilimumab | between week 4 and week 10
  To determine the Maximum Tolerated Dose (MTD), Dose Limiting Toxicity (DLT) andrecommended Phase 2 dose of radiation therapy administered in combination with ipilimumab.

SECONDARY OUTCOMES:
Adverse event profiles | At an average of every four weeks during the treatment phase
  Adverse event profiles
overall survival in patients treated with this combination | At an average of every four weeks during the treatment phase and then every three months during the follow-up phase
  overall survival in patients treated with this combination

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Gustave Roussy Cancer Campus, Villejuif, Val de Marne
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Boutros C, Chaput-Gras N, Lanoy E, Larive A, Mateus C, Routier E, Sun R, Tao YG, Massard C, Bahleda R, Schwob D, Ibrahim N, Khoury Abboud RM, Caramella C, Lancia A, Cassard L, Roy S, Soria JC, Robert C, Deutsch E. Dose escalation phase 1 study of radiotherapy in combination with anti-cytotoxic-T-lymphocyte-associated antigen 4 monoclonal antibody ipilimumab in patients with metastatic melanoma. J Immunother Cancer. 2020 Aug;8(2):e000627. doi: 10.1136/jitc-2020-000627. PMID 32819972
- See also: Related Info — http://igr.fr